CLINICAL TRIAL: NCT02231723
Title: A Phase Ib Clinical Study of BBI608 in Combination With Standard Chemotherapies in Adult Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study of BBI608 in Combination With Standard Chemotherapies in Adult Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-118; BBI608-201PANC (Other: Boston Biomedical, Inc.)
Record Dates: First submitted 2014-08-30; First posted 2014-09-04 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Digestive System Neoplasms; Endocrine Gland Neoplasms; Pancreatic neoplasms; Pancreatic cancer, adult; Pancreatic cancer; Pancreas cancer; Pancreatic diseases; Adenoma, Islet Cell; Carcinoma, Islet Cell; Carcinoma, Pancreatic Ductal; Gemcitabine; Gemzar; Nab-paclitaxel; Paclitaxel; Abraxane; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil; 5-FU; MM-398
MeSH Terms: conditions — Digestive System Neoplasms; Endocrine Gland Neoplasms; Pancreatic Neoplasms; Pancreatic cancer, adult; Pancreatic Diseases; Adenoma, Islet Cell; Carcinoma, Islet Cell; Carcinoma, Pancreatic Ductal | interventions — napabucasin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Paclitaxel; Gemcitabine; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil; irinotecan sucrosofate

ARMS (4):
- A: BBI608 in combination with Gemcitabine and nab-Paclitaxel (Experimental)
  Interventions: Drug: BBI608; Drug: Nab-paclitaxel; Drug: Gemcitabine
- B: BBI608 in combination with modified FOLFIRINOX (Experimental)
  Interventions: Drug: BBI608; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Fluorouracil
- C: BBI608 in combination with FOLFIRI (Experimental)
  Interventions: Drug: BBI608; Drug: Leucovorin; Drug: Irinotecan; Drug: Fluorouracil
- D: BBI608 in combination with MM-398, 5-FU and leucovorin (Experimental)
  Interventions: Drug: BBI608; Drug: Leucovorin; Drug: Fluorouracil; Drug: MM-398

INTERVENTIONS:
Drug: BBI608 — Administered continuously twice daily with doses separated by 12 hours
  Other Names: Napabucasin; BB608; BBI-608
Drug: Nab-paclitaxel — Nab-paclitaxel 125 mg/m^2 I.V. infusion on Days 1, 8, and 15 of every 28-day cycle
  Other Names: Abraxane, nanoparticle albumin-bound paclitaxel, paclitaxel, ABI-007
  Arms: A: BBI608 in combination with Gemcitabine and nab-Paclitaxel
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 I.V. infusion on Days 1, 8, and 15 of every 28-day cycle
  Other Names: Gemzar
  Arms: A: BBI608 in combination with Gemcitabine and nab-Paclitaxel
Drug: Oxaliplatin — Oxaliplatin 85 mg/m^2 I.V. infusion on Days 1 and 15 of every 28-day cycle
  Other Names: Eloxatin
  Arms: B: BBI608 in combination with modified FOLFIRINOX
Drug: Leucovorin — Arm C, D: Leucovorin 400 mg/m^2 I.V. infusion on Days 1 and 15 of every 28-day cycle
  Other Names: Folinic Acid
  Arms: C: BBI608 in combination with FOLFIRI; D: BBI608 in combination with MM-398, 5-FU and leucovorin
Drug: Irinotecan — Arm B: Irinotecan 165 mg/m^2 I.V. infusion on Days 1 and 15 of every 28-day cycle, Arm C: Irinotecan 165 mg/m^2 I.V. infusion on Days 1 and 15 of every 28-day cycle
  Other Names: Camptosar
  Arms: B: BBI608 in combination with modified FOLFIRINOX; C: BBI608 in combination with FOLFIRI
Drug: Fluorouracil — Arm B, D: Fluorouracil 2400 mg/m^2 I.V. infusion on Days 1 and 15 of every 28-day cycle, Arm C: Fluorouracil 400 mg/m^2 I.V. bolus followed by 2400 mg/m^2 I.V. infusion on Days 1 and 15 of every 28-day cycle
  Other Names: 5-FU; Carac; Efudex; Fluoroplex; Adrucil
  Arms: B: BBI608 in combination with modified FOLFIRINOX; C: BBI608 in combination with FOLFIRI; D: BBI608 in combination with MM-398, 5-FU and leucovorin
Drug: MM-398 — MM-398 70 mg/m^2 I.V. infusion on Days 1 and 15 of every 28-day cycle
  Other Names: Onivyde
  Arms: D: BBI608 in combination with MM-398, 5-FU and leucovorin

SUMMARY:
This is an open label, multi-center, multi-arm, dose-escalation study of BBI608 administered in combination with Gemcitabine and nab-Paclitaxel, mFOLFIRINOX, FOLFIRI, or MM-398 with 5-FU and leucovorin.

DETAILED DESCRIPTION:
This is an open label, multi-center, multi-arm, dose-escalation study of BBI608 administered in combination with either Gemcitabine and nab-Paclitaxel, mFOLFIRINOX, FOLFIRI, or MM-398 with 5-FU and leucovorin. A study cycle will consist of daily and continuous oral administration of BBI608 for four weeks (28 days) in combination with Gemcitabine and nab-Paclitaxel, mFOLFIRINOX, FOLFIRI, or MM-398 with 5-FU and leucovorin. Combination treatment will continue in 28 day cycles until disease progression, unacceptable toxicity or another discontinuation criterion is met. BBI608 may be continued post-progression if the patient is obtaining potential clinical benefit, in the opinion of the investigator. If administration of Gemcitabine and/or nab-Paclitaxel, mFOLFIRINOX, FOLFIRI, or MM-398 with 5-FU and leucovorin is discontinued due to chemotherapy backbone-related toxicities, the administration of BBI608 can be continued.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH) - Good Clinical Practice (GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPAA) prior to study-specific screening procedures.
2. Patients must have histologic or cytologic evidence of adenocarcinoma of the pancreas, such as a core tissue biopsy or a surgical resection specimen.
3. Patients must have metastatic disease. Baseline imaging of chest, abdomen and pelvis (CT or MRI) within 21 days prior to initiation of protocol therapy is required.

   1. Patients must have measurable disease as defined by RECIST 1.1.
   2. Patients with locally advanced unresectable pancreatic ductal adenocarcinoma are excluded.
4. Patients enrolling onto Arm A (Gemcitabine and nab-Paclitaxel) or Arm B (mFOLFIRINOX) are allowed to have up to two prior lines of systemic therapy, with adjuvant therapy counted as one line of therapy as long as disease recurrence occurred > 6 months of last dose of therapy. Prior systemic therapy in the metastatic setting is allowed for as long as the therapy contained BBI608 in combination with either Gemcitabine and nab-Paclitaxel or mFOLFIRINOX. Toxicities related to prior therapy must have completely resolved (except for alopecia and anemia), or be deemed irreversible.

   1. Patients who received Gemcitabine-based therapy in an adjuvant setting will be allowed to be enrolled on Arm A of the trial (Gemcitabine with nab-Paclitaxel) as long as their last Gemcitabine administration was at least 6 months prior to the first dose of BBI608.
   2. Patients enrolling onto Arm A (Gemcitabine with nab-Paclitaxel) are allowed to have prior mFOLFIRINOX in combination with BBI608 in the metastatic setting.
   3. Patients enrolling onto Arm B (mFOLFIRINOX) are allowed to have prior Gemcitabine with nab-Paclitaxel in combination with BBI608 in the metastatic setting.
   4. Prior treatment with radiotherapy is allowed.
5. Patients enrolling onto Arm C (FOLFIRI) or Arm D (MM-398 with 5-FU and leucovorin) must have failed one prior line of gemcitabine-based therapy with or without BBI608 in the metastatic setting. No additional lines of therapy in the metastatic setting are allowed. Prior adjuvant therapy with gemcitabine is allowed as long as disease recurrence occurred > 6 months of last dose of therapy. Toxicities related to prior therapy must have completely resolved (except for alopecia and anemia), or be deemed irreversible. Prior treatment with radiotherapy is allowed.
6. ≥ 18 years of age.
7. Patients must have an ECOG Performance Status ≤ 1.
8. Male or female patients of child-producing potential agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI608 dose.
9. Females of childbearing potential have a negative serum pregnancy test (preceding 72 hours of first day of BBI608 treatment).
10. Patients with biliary or gastro-duodenal obstruction must have drainage or surgical bypass prior to starting chemotherapy.
11. Significant or symptomatic amount of ascites should be drained prior to first dose of BBI608.
12. Patients on Warfarin/Dabigatran/Rivaroxaban anticoagulation may be enrolled for as long as they undergo weekly INR checks for the first 2 months of therapy.

    a. Patients who switch to low molecular weight heparin may be enrolled and weekly INR labs are not mandated for these patients.
13. Aspartate transaminase (AST) level ≤ 2.5 x upper limit of normal (ULN) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN). For patients with liver metastases, AST ≤ 5 ULN, and AST ≤ 5 ULN may be enrolled if agreed upon by the investigator and medical monitor for the sponsor.
14. Patients must have a total bilirubin level ≤ 1.5 x ULN (≤ 2 x ULN if it is non-rising for a period of 10 days prior to initiation of therapy).
15. Creatinine level < 1.0 x ULN or creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above or below the institutional normal (as determined by Cockcroft-Gault equation). For patients with a Body Mass Index (BMI) > 30 kg/m^2, lean body weight should be used to calculate the GFR.
16. Hemoglobin (Hgb) ≥ 9 g/dl
17. Absolute neutrophil count ≥ 1.5 x 10^9/L
18. Platelets ≥ 100 x 10^9/L
19. Acceptable coagulation studies as demonstrated by prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits (+/-15%).
20. Patient has no clinically significant abnormalities on urinalysis results.
21. Life expectancy estimated at ≥ 3 months.

Exclusion Criteria:

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within 14 days of the first dose of BBI608, except for BBI608 for which a washout period is not required.

   1. Patients may begin BBI608 on a date determined by the investigator and medical monitor for the sponsor after a minimum of 14 days since last receiving anti-cancer treatment which did not include BBI608, provided that all treatment-related adverse events have resolved or have been deemed irreversible (except for alopecia).
   2. Patients who previously received BBI608 for treatment of PDAC on the BBI608-118 (BBI608-201PANC) study may continue with BBI608 in monotherapy between discontinuation of the first chemotherapy backbone and start of the second chemotherapy backbone. Patients may begin chemotherapy backbone on a date determined by the investigator and medical monitor for the sponsor after a minimum of 14 days and a maximum of 30 days since last receiving anti-cancer treatment which included BBI608, provided that all treatment-related adverse events have resolved or have been deemed irreversible (except for alopecia).
2. Patients with neuroendocrine neoplasms will be excluded.
3. Major surgery, other than diagnostic surgery (e.g., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to first dose.
4. Any brain metastases including leptomeningeal metastases, are excluded, even if treated and stable.
5. History of posterior reversible encephalopathy syndrome.
6. Neurosensory neuropathy ≥ grade 2 at baseline.
7. Pregnant or breastfeeding.
8. Significant gastrointestinal disorder(s) that would, in the opinion of the Principal Investigator, prevent absorption of an orally available agent (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection and small intestinal resection).
9. Unable or unwilling to swallow BBI608 capsules daily.
10. Uncontrolled chronic diarrhea ≥ grade 2 at baseline.
11. Uncontrolled intercurrent illness including, but not limited to uncontrolled active infection (including bacterial, viral or fungal requiring systemic therapy), clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
12. Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
13. History of other active malignancies.
14. Enrollment on any additional investigational agent study. Enrollment on concurrent observational study is allowed following consultation with the Sponsor.
15. Patients planning to take a vacation for 7 or more consecutive days during the course of the study.
16. For patients enrolling onto Arm A (Gemcitabine with nab-Paclitaxel)

    a. Known hypersensitivity to Gemcitabine or taxanes. i. Patients with history of Gemcitabine toxicity in the adjuvant setting requiring more than 1 dose level reduction are excluded.

    b. Significant cardiac disease, including the following: unstable angina, New York Heart Association class III-IV congestive heart failure, myocardial infarction within six months prior to study enrollment.

    c. History of hemolytic-uremic syndrome. d. History of posterior reversible encephalopathy syndrome. e. Known infection with Human Immunodeficiency Virus (HIV), and/or active infection with hepatitis B, or hepatitis C.

    f. History of active Peripheral Artery Disease (treated peripheral artery disease that is stable for at least 6 months is allowed).
17. For patients enrolling onto Arm B (mFOLFIRINOX) or Arm C (FOLFIRI)

    1. Known hypersensitivity to 5-fluorouracil/leucovorin
    2. Known dihydropyrimidine dehydrogenase (DPD) deficiency
    3. Known hypersensitivity to oxaliplatin or other platinum containing compounds
    4. Known hypersensitivity to irinotecan
    5. Uncontrolled seizure disorder, active neurological disease, or known CNS disease.
    6. Known Gilbert's syndrome
    7. Significant cardiac disease, including the following: unstable angina, New York Heart Association class II-IV congestive heart failure, myocardial infarction within six months prior to study enrollment.
18. For patients enrolling onto Arm D (MM-398 with 5-FU and leucovorin)

    1. Prior irinotecan treatment
    2. Arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) < 6 months prior to enrollment
    3. Known hypersensitivity to any of the components of MM-398, other liposomal products, fluoropyrimidines or leucovorin
    4. Known dihydropyrimidine dehydrogenase (DPD) deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-08; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Safety by reporting the adverse events and serious adverse events | 6 months
Determination of the Recommended Phase 2 Dose by assessing dose-limiting toxicities (DLTs) | 3 months

SECONDARY OUTCOMES:
Assess the preliminary anti-tumor activity of BBI608 when administered in combination with standard chemotherapies by performing tumor assessments every 8 weeks | 6 months
Assess the preliminary anti-tumor activity of BBI608 when administered in combination with standard chemotherapies by performing serum CA 19-9 level measurement | 6 months
  Assess the preliminary anti-tumor activity of BBI608 when administered in combination with standard chemotherapies in adult patients with metastatic pancreatic adenocarcinoma by performing serum carbohydrate antigen 19-9 (CA 19-9) level measurement every 4 weeks
Assess pharmacokinetic profile of BBI608 when administered in combination with standard chemotherapies | On Day 1 and Day 15 of the first cycle prior to dosing and 1, 2, 3, 3.5, 4, 5, 5.5, 7, 8, 9, 10, 11 and 24 hours after first dose
  Blood sampling to assess the pharmacokinetic profile (Area under the curve) of BBI608.
Assess pharmacodynamic activity of BBI608 when administered in combination with standard chemotherapies | During the first 28 days of treatment
  Tumor Biopsy to provide information of the biomarkers by histopathology and Cancer Stem Cell assays.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - SAT&BC, San Antonio, Texas
  - Virginia Oncology Associates, Norfolk, Virginia